CLINICAL TRIAL: NCT00526591
Title: Randomized Phase II Study of Two Different Doses of RAD-001 (Everolimus) as Neo-Adjuvant Therapy in Patients With Localized Prostate Cancer
Brief Title: Everolimus in Treating Patients With Newly Diagnosed Localized Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Jorge A. Garcia, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Jorge A. Garcia, MD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE21806; P30CA043703 (NIH); CASE-21806 (Other: Case Comprehensive Cancer Center); CASE-21806-CC256 (Other: Cancer Center IRB)
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-dose Everolimus Cohort (Experimental): 5mg Everolimus daily continuously for 8 weeks and conventional surgery
  Interventions: Drug: Everolimus; Procedure: conventional surgery
- High-dose Everolimus Cohort (Active Comparator): 10mg Everolimus daily continuously for 8 weeks and conventional surgery
  Interventions: Drug: Everolimus; Procedure: conventional surgery

INTERVENTIONS:
Drug: Everolimus — Patients will receive arm-specific dosage of Everolimus daily continuously for 8 week
  Other Names: RAD-001
Procedure: conventional surgery — Radical prostatectomy with bilateral pelvic lymphadenectomy will be performed within 10 days of the completion of week 8 on RAD-001 (Everolimus).

SUMMARY:
RATIONALE: Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving everolimus before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This randomized phase II trial is studying the side effects and how well everolimus works in treating patients with newly diagnosed localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the clinical effects of everolimus, in terms of pathologic response (i.e., histologic P0, margin status, or capsular penetration) and surgical outcome, in patients with newly diagnosed localized prostate cancer treated with two different doses of everolimus prior to radical prostatectomy.
* To evaluate the safety and tolerability of this drug in these patients.

Secondary

* To determine the effect of this drug on prostate-specific antigen (PSA) levels in these patients.
* To determine the effect of this drug on levels of expression of PTEN, Akt, phospho-mTOR (i.e., Se2448), phospho-p70 S6 kinase (i.e., Thre389), phospho-Smad3 (i.e., Ser433/435), phospho-Smads 1/5 (i.e., Ser463/465), AR, and TUNEL in these patients.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive low-dose oral everolimus once daily for up to 8 weeks in the absence of unacceptable toxicity.
* Arm II: Patients receive high-dose oral everolimus once daily for up to 8 weeks in the absence of unacceptable toxicity.

Within 7 days after the last dose of everolimus, all patients undergo radical prostatectomy with bilateral pelvic lymphadenectomy.

Tumor biopsy specimens acquired prior to treatment and prostate tumor tissue acquired at the time of radical prostatectomy are evaluated for biomarker correlative studies. Tissue samples are assessed by immunohistochemistry (IHC) and tissue microarray analysis for expression of cellular and molecular biomarkers (i.e., p-S6, p-4E-BP1, and p-Akt) that correlate with response. Prostatectomy specimens are also assessed by pathologic analysis for histopathologic response (i.e., pathologic stage, Gleason score, margin status, and tumor size).

After completion of study therapy, patients are followed at 6 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed newly diagnosed, localized adenocarcinoma of the prostate, meeting any of the following criteria:

  * Clinical stage T2a, T2b, T2c, or T3 disease (any grade or PSA)
  * Gleason score 7 (4+3 only) or ≥ 8 (any stage or PSA)
  * Serum PSA ≥ 10 ng/dL (any grade or stage)
  * Any stage, PSA, or Gleason score AND ≥ 35% chance of biochemical failure at 5 years based on Kattan's nomogram
* Recommended for radical prostatectomy
* Normal testosterone level
* No pure neuroendocrine or small cell prostate cancer
* No metastatic disease by CT scan, MRI, bone scan, or X-ray
* No clinical evidence of CNS metastases

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status (PS) 0-1 or Karnofsky PS 70-100%
* ANC ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Hemoglobin ≥ 8 g/dL
* AST and ALT ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* Creatinine ≤ 1.5 times ULN
* PT/PTT normal (no anticoagulants)
* No active unresolved infection
* No known HIV positivity
* Fertile patients must use effective contraception during and for 6 months after completion of study therapy

Exclusion criteria:

* Known hypersensitivity to everolimus or other rapamycins (e.g., sirolimus or temsirolimus) or to its excipients
* Gastrointestinal (GI) disease, condition, or symptoms that may significantly impair GI function and alter the absorption of everolimus, including any of the following:

  * Ulcerative disease
  * Uncontrolled nausea
  * Vomiting
  * Diarrhea
  * Malabsorption syndrome
* Other active malignancy or malignancy at ≥ 30% risk for relapse after completion of therapy, except nonmelanoma skin cancer
* Uncontrolled concurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection (e.g., bacterial, viral or fungal)
  * Severely impaired lung function
  * Uncontrolled diabetes (fasting serum glucose > 1.5 times ULN)
  * Liver disease (e.g., cirrhosis, chronic active hepatitis, or chronic persistent hepatitis)
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
* Psychiatric illness or social situation that would limit study compliance
* Any underlying medical condition which, in the principal investigator's opinion, will make the administration of everolimus hazardous OR obscure the interpretation of adverse events

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since major surgery
* More than 3 months since finasteride
* No prior or concurrent radiotherapy to the prostate gland or pelvis
* No prior hormones (e.g., luteinizing hormone-releasing hormone [LHRH] agonists, LHRH antagonists, or antiandrogens [e.g., bicalutamide, flutamide, or nilutamide]) and/or PC-SPES (or PC-x product) or estrogen-containing nutraceuticals
* No prior rapamycin mTOR inhibitor
* No prior small bowel resection that may significantly impair GI function and alter the absorption of everolimus
* No prior or concurrent immunotherapy, chemotherapy, or other investigational therapy for prostate cancer
* No other concurrent investigational or commercial agents
* No other concurrent anticancer agents
* No concurrent, chronic treatment with systemic steroids (except inhaled or topical steroids) or another immunosuppressive agent
* No concurrent live vaccines
* No concurrent strong inhibitors or inducers of the isoenzyme CYP3A administered as systemic therapy

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-09; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge A. Garcia, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Koshkin VS, Mir MC, Barata P, Gul A, Gupta R, Stephenson AJ, Kaouk J, Berglund R, Magi-Galluzzi C, Klein EA, Dreicer R, Garcia JA. Randomized phase II trial of neoadjuvant everolimus in patients with high-risk localized prostate cancer. Invest New Drugs. 2019 Jun;37(3):559-566. doi: 10.1007/s10637-019-00778-4. Epub 2019 Apr 30. PMID 31037562

RESULTS

PARTICIPANT FLOW:
Groups:
- Low-dose Cohort: Patients will receive 5.0mg P.O. daily continuously for 8 weeks
  everolimus: Low-dose Cohort: Patients will receive 5.0mg P.O. daily continuously for 8 weeks; High-dose Cohort: Patients will receive 10mg P.O. daily continuously for 8 weeks
  conventional surgery: Radical prostatectomy with bilateral pelvic lymphadenectomy will be performed within 10 days of the completion of week 8 on RAD-001 (Everolimus).
- High-dose Cohort: Patients will receive 10mg P.O. daily continuously for 8 weeks
  everolimus: Low-dose Cohort: Patients will receive 5.0mg P.O. daily continuously for 8 weeks; High-dose Cohort: Patients will receive 10mg P.O. daily continuously for 8 weeks
  conventional surgery: Radical prostatectomy with bilateral pelvic lymphadenectomy will be performed within 10 days of the completion of week 8 on RAD-001 (Everolimus).
Period: Overall Study
Arm/Group | Low-dose Cohort | High-dose Cohort
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-dose Cohort | High-dose Cohort | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (7.9) | 59 (4.5) | 59 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 9 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Are P0 (i.e., no Clinically Detectable Tumor in the Pathologic Specimen) at Surgery
Description: Specimens are fixed in formalin for 24 hours.Specimens are the cut at 3 mm intervals perpendicular to the rectal surface and the sections are examined grossly and microscopically on routine Hematoxylin and Eosin stain (H&E) (pathologic complete response or P0) will be defined as responders.
Time Frame: After 8 weeks of therapy at the time of prostatectomy
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Low-dose Cohort | High-dose Cohort
Number analyzed (Participants) | 8 | 9
participants | 0 | 0

2. Primary Outcome: Toxicity Profile of Each Dose (Number of Patients With Worst Grade Toxicity)
Description: Toxicity will be assessed using the NIH-NCI Common Terminology Criteria for Adverse Events, version 3.0 (CTCAEv3.0)
Time Frame: at daily dose for 8 weeks
Population: intention to treat
Measure: Number; unit: participants
Arm/Group | Low-dose Cohort | High-dose Cohort
Number analyzed (Participants) | 8 | 9
participants
  Patients with Grade 3 toxicity | 2 | 1
  Patients with Grade 4 toxicity | 0 | 0

3. Secondary Outcome: Change in PSA
Description: Time-to-event data, such as change in PSA will be summarized using the method of Kaplan and Meier.
Time Frame: Up to 16 weeks after start of study
Population: One patient in the high dose cohort was not analyzed for change in PSA because they withdrew early due to progressive disease
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | High-dose Cohort | Low-dose Cohort
Number analyzed (Participants) | 8 | 8
ng/mL | 3.5 [-0.8 to 21.6] | 3.04 [-4.2 to 58.4]

4. Other Pre Specified Outcome: Effect of Treatment on Biological and Molecular Markers
Description: Immunohistochemical Staining of Cellular and Molecular Markers in Prostate Tumor Tissue
Time Frame: After 8 weeks of therapy
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: At daily dose for 8 weeks
Arm/Group | Low-dose Cohort | High-dose Cohort
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/9
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose Cohort (N=8) | High-dose Cohort (N=9)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose Cohort (N=8) | High-dose Cohort (N=9)
Anorexia (Metabolism and nutrition disorders) | 1 (2) | 3 (3)
Aspartate aminotransferase (Investigations) | 4 (4) | 2 (2)
hemoglobin (Investigations) | 1 (1) | 5 (5)
Cholesterol high (Investigations) | 5 (7) | 4 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Creatinine (Investigations) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Sensation of coldness (General disorders) | 1 (1) | 0 (0)
dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Furuncle (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dry eye syndrome (Eye disorders) | 2 (2) | 0 (0)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Edema: limb (General disorders) | 1 (1) | 3 (5)
Erectile dysfunction (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5 (6) | 3 (5)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 5 (7) | 2 (2)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incontinence, urinary (Renal and urinary disorders) | 7 (8) | 4 (4)
infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Stabbing rectal pain Infection with normal ANC (Infections and infestations) | 1 (1) | 0 (0)
insominia (Psychiatric disorders) | 1 (1) | 0 (0)
libido (Psychiatric disorders) | 1 (1) | 0 (0)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 5 (11) | 7 (12)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pain - Back (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain - Chest/thorax NOS (General disorders) | 2 (2) | 0 (0)
Pain - Head/headache (Nervous system disorders) | 3 (3) | 3 (4)
Pain broken tooth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (2) | 5 (5)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
bronchial mucous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 3 (5) | 5 (5)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 1 (1)
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 0 (0) | 1 (1)
Bicarbonate, serum-low (Investigations) | 0 (0) | 1 (1)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hair Color change (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flu-like syndrome (General disorders) | 0 (0) | 1 (1)
Hot flashes/flushes (Vascular disorders) | 0 (0) | 1 (1)
Infection, lower lip (Infections and infestations) | 0 (0) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (5)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 0 (0) | 2 (2)
Pain, left heel (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain, left groin (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pain and burning while urinating (Renal and urinary disorders) | 0 (0) | 1 (1)
Pain at surgery site (Investigations) | 0 (0) | 1 (1)
pain,left groin (Reproductive system and breast disorders) | 0 (0) | 1 (1)
pain/rectal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain, throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Platelets (Investigations) | 0 (0) | 5 (6)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
nocturia (Renal and urinary disorders) | 0 (0) | 3 (3)
Rigors/chills (General disorders) | 0 (0) | 1 (1)
Sweating (diaphoresis) (General disorders) | 0 (0) | 1 (1)
Taste alteration (dysgeusia) (Nervous system disorders) | 0 (0) | 2 (2)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes